CLINICAL TRIAL: NCT05122975
Title: Treatment of Catecholaminergic Polymorphic Ventricular Tachycardia Type 1 (CPVT1)
Brief Title: Treatment of an Inherited Ventricular Arrhythmia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to challenges in recruiting patients.
Sponsor: RyCarma Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL2-210-01; 1R01FD007279-01 (FDA)
Record Dates: First submitted 2021-10-22; First posted 2021-11-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Catecholaminergic Polymorphic Ventricular Tachycardia Type 1
Keywords: Ventricular Arrhythmia; Calcium; Ryanodine Receptor 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: S48168 and exact matching placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S48168 (ARM210) once daily for 28 days (Experimental): Oral dose of S48168 (ARM210) once daily on top of standard of care regimen for 28 days.
  Interventions: Drug: S48168 (ARM210)
- Matching Placebo once daily for 28 days (Placebo Comparator): Oral dose of placebo once daily on top of standard of care regimen for 28 days.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: S48168 (ARM210) — Ryanodine Receptor modulator
  Arms: S48168 (ARM210) once daily for 28 days
Drug: Matching Placebo — Placebo of same size and consistency as S48168 (ARM210)
  Arms: Matching Placebo once daily for 28 days

SUMMARY:
The goal of the proposed project is to determine the safety and tolerability as well as the preliminary efficacy of a novel small molecule drug, S48168 (ARM210), for the treatment of Catecholaminergic Polymorphic Ventricular Tachycardia (CPVT1). This disease is associated with fatal changes in heart rhythms leading to sudden death with exercise or excessive excitement. It is due to mutations in the Ryanodine Receptor calcium release channel, which cause leaky channels leading to the disease. S48168 (ARM210) repairs these leaky channels and can be a disease-modifying therapy restoring normal function to the channels. This result would allow patients with CPVT to live normal, active lives. Funding Source- FDA OOPD.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following conditions to be eligible for enrollment into the study:

1. Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
2. Participants who are willing and able to comply with scheduled visits, study drug administration plan, study restrictions, and study procedures.
3. Participants have a confirmed genetic diagnosis of CPVT1 and supporting clinical phenotype, including residual ventricular ectopy (a complexity score ≥ 2; requiring at minimum the presence of PVCs in bigeminy on exercise stress test) on a stable (at least 1 month) standard-of-care, CPVT1-directed treatment regimen as decided by their CPVT treating physician.
4. Have a body mass index (BMI) ≤ 36 kg/m2 (inclusive) at screening.
5. Male participants agree to not donate sperm from the first day of dosing of study drug until 5 half-lives plus 90 days (approximately 94 days) after the last dose of study drug.

   Female participants:

   eligible to participate if she is not pregnant or breastfeeding, and uses one of the following highly effective birth control methods (from the first dose until 5 half-lives plus 90 days (approximately 94 days):
   * Prescribed hormonal oral contraceptives, vaginal ring, or transdermal patch.
   * Intrauterine device (IUD).
   * Intrauterine hormone-releasing system (IUS).
   * Depot/implantable hormone (e.g., Depo-Provera®, Implanon).
   * Bilateral tubal occlusion/ligation.
   * Sexual abstinence.
   * Refraining from heterosexual intercourse during the entire period of risk associated with the study requirements.
   * If the participant decides to become sexually active during the study, then one of the highly effective birth control methods must be used.

   OR

   Is a woman of non-childbearing potential; defined by at least 1 of the following criteria:
   * Postmenopausal defined as 12 months of spontaneous amenorrhea without a medical cause and follicle stimulating hormone (FSH) serum level > 40 mIU/mL without the use of hormonal supplementation. Appropriated documentation of FSH levels is required.
   * Surgically sterile by hysterectomy and/or bilateral oophorectomy with appropriate documentation of surgical procedure.
   * Has a congenital condition resulting in no uterus.
6. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
7. Daily use of medicines and dietary supplements need to be approved by the PI and Sponsor, or a drug/supplement-dependent wash-out prior to inclusion.

Exclusion Criteria:

The presence of any of the following conditions will exclude a participant from study enrollment:

1. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose of study drug.
2. History or presence of hypersensitivity or idiosyncratic reaction to the study drug, related compounds, or inactive ingredients.
3. ALT or AST levels three times above the upper limits of normal (ULN) at screening (isolated elevations of total bilirubin < 2 X ULN with direct bilirubin below the ULN will be included). A recheck for confirmation is allowed.
4. History of documented, EEG-confirmed epileptic seizures.
5. History of cancer (malignancy). Exceptions: (1) Subjects with adequately treated non-melanomatous carcinoma or carcinoma in situ of the cervix may participate in the trial; (2) Subjects with other malignancies who have been successfully treated > 10 years prior to the screening where in the judgment of the investigator has revealed no evidence of recurrence from the time of treatment through the time of the screening except those identified at the beginning of the exclusion criterion; or (3) Subjects who in the opinion of the investigator are highly unlikely to sustain a recurrence for the duration of the trial.
6. Currently has uncontrolled diabetes defined as HbA1c > 7% at screening visit or diabetic neuropathy.
7. Estimated creatinine clearance < 40mL/minute at screening visit.
8. Clinically significant abnormality on their screening and/or prior to first dosing resting ECG, other than hypertensive related, or heart failure (ejection fraction < 30%) or other clinically significant structural heart disease.
9. History of myocardial infarction in the last five years, or evidence of congestive heart failure.
10. Ongoing medical condition that is deemed by the PI to interfere with the conduct or assessments of the study or safety of the subject.
11. Unable to refrain from or anticipates the use of:

    * Any non-approved medicines (prescribed standard-of-care for CPVT is approved) and/or dietary supplements beginning 14 days prior to the first dose of study drug and throughout the study. Thyroid hormone replacement medication may be permitted if subject has been on same stable dose for the last 3 months prior to the first dose of study drug.
    * Any drugs known to be significant inducers or inhibitors of CYP2C8 enzymes for 28 days prior to the first dose of study drug and throughout the study. Is currently taking any drug which raises gastric pH, including proton pump inhibitors or H2 antagonists. Antacids may be used if taken at night.
12. Participation in clinical trials for other therapeutic investigational drugs simultaneously or within the 4 weeks prior to the first dose of study drug.
13. Plasma donation within 7 days prior to the first dose of study drug.
14. Donation of blood or significant blood loss within 56 days prior to the first dose of study drug.
15. Is mentally or legally incapacitated at the time of screening visit.
16. Is unable to take orally administered tablets.
17. Is an immediate family member of the Sponsor or employee of the clinical site or may consent under duress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
The effect of S48168 (ARM210) treatment on the amount and complexity of exercise-• Change in ectopy score from baseline to Day 28 versus placebo (pre-dose Period 1 baseline to Day 28 Period 1 versus Day 28 Period 2 | 28 days
  Analysis of ECG recordings during exercise testing examining for abnormal beats occurring with exercise, such as premature ventricular contractions (PVCs). The scale is as follows:
  Ectopy Scoring Scale (0-4)
  No ectopy 0
  Isolated PVCs 1
  Bigeminy 2
  Couplets 3
  Non-sustained VT 4
  van der Werf, C., et al. (2011). "Flecainide therapy reduces exercise-induced ventricular arrhythmias in patients with catecholaminergic polymorphic ventricular tachycardia." J Am Coll Cardiol 57(22): 2244-2254.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 28 days
  The number and severity of adverse events that can be related to treatment with S48168 (ARM210)

OTHER OUTCOMES:
The pharmacokinetics (PK) of a 28-day administration of S48168 (ARM210) in patients | 28 days
  Day one and day 28 maximal plasma concentration (Cmax)
Total Plasma Drug Exposure of a 28-day administration of S48168 (ARM210) in patients | 28 days
  Measurement of the area under the curve (AUC) at day 1 and day 28 in plasma
Evaluation of a novel expanded ectopy scale in exercise stress tests which qualifies both the ectopy and the heart rate at which it occurs. | 28 days
  Expanded novel ectopy scale No ectopy 0 points PVCs only 1 point Bigeminy 2 points Couplets 5 points Non-sustained VT 10 points Add 5 points for ectopy onset at heart rate <=120 bpm; 3 points for ectopy onset at heart rate > 120 but <= 150 bpm; 1 point for ectopy onset at heart rate > 150 bpm
Evaluation of heart rhythm throughout treatment periods | 28 days
  Using a wearable cardiac monitoring device continuously throughout the treatment periods to determine frequency of abnormal beats including PVCs, bigeminy and couplets in the active and placebo treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Ackerman, MD PhD, Principal Investigator — Mayo Clinic
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Amsterdam University Medical Center, Amsterdam-Zuidoost, Netherlands

IPD SHARING:
Plan to Share IPD: No